CLINICAL TRIAL: NCT07080606
Title: Brief Exposure and Exercise Therapy for Post Traumatic Stress Disorder (PTSD)
Brief Title: Brief Exposure and Exercise for PTSD.
Acronym: BEE for PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Troy Hubert (Other)
Responsible Party: Sponsor-Investigator, Troy Hubert, Graduate Research Assistant, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101765
Record Dates: First submitted 2025-07-01; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: PTSD - Post Traumatic Stress Disorder
Keywords: PTSD; Exercise; Exposure Therapy
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic; Motor Activity | interventions — Exercise; Implosive Therapy

STUDY DESIGN:
Intervention Model Description: Acceptability and Feasibility using a Single Case Experimental Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Brief exposure therapy and exercise 3 week (Experimental): Participants are randomized into the 3 week baseline condition before receiving the exposure therapy and exercise intervention.
  Interventions: Behavioral: Brief exposure therapy and exercise
- Brief exposure therapy and exercise 5 week (Experimental): Participants are randomized into the 5 week baseline condition before receiving the exposure therapy and exercise intervention.
  Interventions: Behavioral: Brief exposure therapy and exercise
- Brief exposure therapy and exercise 4 week (Experimental): Participants are randomized into the 4 week baseline condition before receiving the exposure therapy and exercise intervention.
  Interventions: Behavioral: Brief exposure therapy and exercise

INTERVENTIONS:
Behavioral: Brief exposure therapy and exercise — Treatment provided in this study includes an open label brief imaginal exposure therapy for Post Traumatic Stress Disorder (PTSD) and moderate intensity aerobic exercise (i.e., 70-75% max heart rate). Participants all receive 30 minutes of psychotherapy and 25 minutes of exercise.
  Other Names: Imaginal Exposure

SUMMARY:
The goal of this clinical trial is to learn if 8 sessions of brief exposure and exercise therapy works to treat Post Traumatic Stress Disorder (PTSD) in adults. This study will also learn if participants think brief exposure and exercise therapy is a good and doable treatment. and The main questions it aims to answer are:

* Do participants find brief exposure and exercise an acceptable and feasible means of treatment for PTSD?
* Does brief exposure and exercise decreases of the severity of PTSD symptoms?

Participants will:

* Complete weekly questionnaires for 10-14 weeks.
* Attend 8 twice weekly exposure therapy and exercise sessions for 4 weeks.

DETAILED DESCRIPTION:
A community sample (n=6) of adults with PTSD will receive eight sessions of standardized brief exposure therapy with six sessions of imaginal exposures and aerobic exercise. This clinical trial will be the first study demonstrate the effectiveness of an exposure-only therapy and exercise treatment by isolating and targeting safety learning using imaginal exposures. This approach will address gaps in the literature by demonstrating treatment effectiveness, mechanistic engagement, and patients' perceptions of a brief imaginal exposure treatment combined with aerobic exercise. Addressing these gaps through a preliminary clinical trial that establishes feasibility and treatment effectiveness is a necessary first step before exerting substantial time and money on a large-scale clinical trial.

Aligned with an experimental therapeutics approach, the proposed study will take advantage of single-case experimental design (SCED) to explore changes in PTSD symptom severity and exposure therapy mechanisms (i.e., belief change, experiential avoidance, and emotional intensity) within each participant. SCEDs are parsimonious research designs that are ideal for investigating mechanisms and the effectiveness of interventions. SCEDs use each subject as their own control, resulting in high internal validity and the ability to examine effect sizes across subjects.

Upon referral to the study, participants will complete a brief battery of self-report questionnaires to screen for eligibility. Likely eligible participants, determined by the prescreening, will be given a link to schedule an intake with PI or other graduate student research personnel to complete informed consent and assessments to evaluate inclusion/exclusion criteria. Eligible participants will then be randomized to either a 3, 4 or 5 week baseline period, where participants will complete weekly self-report questionnaires to assess PTSD symptoms and exposure therapy mechanisms. Participants fill out a questionnaire battery before, during, and after treatment resulting in a total of 10-14 weeks of self-report assessments. After the baseline assessment phase, participants will complete the first session of PE, which focuses on psychoeducation and treatment planning, six sessions of imaginal exposures and exercise, and a final PE session discussing relapse prevention and future directions. During the six imaginal exposure sessions (sessions 2-7), participants will complete 20 minutes of imaginal exposure to traumatic memories, 10 minutes of emotional processing, and then 20 minutes of moderate-intensity exercise (i.e., 70-75% of MHR) on a stationary bike with 3 minutes of warmup and 2 minutes of cool-down. Proximal measures for exposure mechanisms will be assessed during treatment sessions (e.g., subjective units of distress) to align with distal measures of exposure therapy, which are assessed in the weekly self-report batteries. Following completion of the treatment, participants will be asked to provide satisfaction ratings on the treatment.

PTSD symptom severity will be assessed weekly to investigate treatment efficacy (Aim 1). Acceptability will be evaluated using a self report patient satisfaction questionnaires (Aim 2). Adherence to the treatment protocol will be used to characterize feasibility (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent and are willing to participate in therapy sessions twice weekly, which include moderate-intensity aerobic exercise.
* Participants must be adults aged 18-64 meeting the criteria for PTSD within the past month, who are not currently receiving treatment from other psychotherapy or are on unstable psychiatric medication (i.e., less than four weeks of psychiatric medication).
* Participants should be able to engage in 25 minutes of moderate-intensity aerobic exercise (i.e., 70-75% of max heart rate).
* Participants must be able to speak and read English fluently to participate in the current study.

Exclusion Criteria:

* Participants who endorse health condition(s) that would prevent moderate exercise.
* Participants who endorse (i.e., "yes") any items on the Physical Activity Readiness Questionnaire (PARQ) that is not controlled or managed.
* Participants with any injuries to the lower extremities that may hinder riding an exercise bicycle.
* Psychiatric exclusion criteria include recent (within the past three months) severe use disorder(s), high risk for suicide (i.e., plan, intent, or recent attempt), mania, or psychotic symptoms unrelated to PTSD symptoms.
* Participants currently seeking or undergoing any other trauma-focused psychotherapy treatment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD Checklist for DSM-5 (PCL-5) | Up to 15 weeks.
  The PCL-5 is a 20-item self-report questionnaire used to assess PTSD symptom severity. Each of the 20 PCL-5 items corresponds to symptoms of PTSD in the DSM-5. Items are rated on a Likert scale from 0 (not at all) to 4 (extremely) based upon how bothered participants are by each symptom. Items on the PCL-5 are summed, resulting in a total score of PTSD symptom severity from 0-80. Scores >30 indicate probable PTSD.
Patient Satisfaction Questionnaire Scores | Once at end of treatment (up to 9 weeks).
  Acceptability will be assessed using a patient satisfaction questionnaire. The 5 Items on the patient satisfaction questionnaire are rated on a 4 likert scale with higher scores on the indicating better perceptions of treatment. Total satisfaction of treatment can be obtained by averaging scores across the 5 items.
Feasibility of the intervention | 4 weeks of treatment following the 3-to 5-week baseline.
  Feasibility will be analyzed by examining adherence to the treatment protocol checklist. An average score of 80% treatment adherence for all participants will be used as a threshold to define the feasibility of this intervention.

SECONDARY OUTCOMES:
Changes in Brief Experiential Avoidance Questionnaire | Up to 15 weeks
  The brief experiential avoidance questionnaire (BEAQ) is a 15-item questionnaire that assesses avoidance of unwanted internal experiences, such as uncomfortable emotions, thoughts, memories, or sensations. The BEAQ has a range of 15-90, with high scores indicating more experiential avoidance.
Changes in the posttraumatic cognitions inventory-9 (PTCI-9) | Up to 15 weeks.
  The PTCI-9 is a 9-item self-report that assesses posttraumatic cognitions following traumatic experiences. Items on the PTCI-9 are scored on a likert scale from 0 (Strongly Disagree) to 7 (Strongly Agree) and are averaged for a total score ranging from 0-7. Higher scores indicate higher levels of post-traumatic cognitions.
Changes in the positive and negative valence affect schedule (PANAS) | Up to 15 weeks.
  The negative affect subscale of the PANAS will be anchored to participants' Criterion A (i.e., index) trauma and used to assess for negative affect related to participants' PTSD over the past week. The negative affect subscale is a 10-item self-report measure rated on a Likert scale from 1 (Very slightly or not at all) to 5 (Extremely), with summed scores ranging from 10 to 50. Higher scores indicate higher levels of negative emotions and affect.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Burris, Ph.D., Study Director — University of Kentucky; Shannon Sauer-Zavala, Ph.D., Study Director — University of Kentucky; Troy J.J. Hubert, M.S., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data for participants will be shared. This includes data used for primary analysis, a data dictionary defining all variables, a data analytic plan, and R code used for analysis. All IPD will be hosted on OSF and Github.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: IPD and supporting information will be released before the completion of the first participant and stored after the completion of the study. Data analytic plan and analytic code will be stored on github indefinitely.
Access Criteria: The full de-identified dataset will be released by PI to other researchers upon request. The small de-identified dataset of variables used for primary analysis, the data dictionary, data analytic plan, and the R analytic code will be stored on Github and OSF.
URL: https://github.com/Troy-Hubert/brief-exposure-and-exercise

REFERENCES:
- See also: A Github repository hosting data, analytic plan, and analytic R code. — https://github.com/Troy-Hubert/brief-exposure-and-exercise